CLINICAL TRIAL: NCT00730639
Title: A Phase 1, Open-Label, Multicenter, Multidose, Dose Escalation Study of BMS-936558 (Nivolumab) in Subjects With Selected Advanced or Recurrent Malignancies
Brief Title: A Phase 1 Study of Nivolumab (BMS-936558) in Subjects With Advanced or Recurrent Malignancies
Acronym: MDX1106-03
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-003; MDX1106-03 (Other: BMS)
Record Dates: First submitted 2008-08-04; First posted 2008-08-08 (Estimated); Results first posted 2016-04-15 (Estimated); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Metastatic Castration-resistant Prostrate Cancer; Renal Cell Carcinoma; Metastatic Melanoma; Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Melanoma; Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Melanoma - BMS-936558 (MDX-1106) (Experimental)
  Interventions: Biological: BMS-936558 (MDX-1106)
- RCC - BMS-936558 (MDX-1106) (Experimental)
  Interventions: Biological: BMS-936558 (MDX-1106)
- mCRPC - BMS-936558 (MDX-1106) (Experimental)
  Interventions: Biological: BMS-936558 (MDX-1106)
- NSCLC - BMS-936558 (MDX-1106) (Experimental)
  Interventions: Biological: BMS-936558 (MDX-1106)
- CRC - BMS-936558 (MDX-1106) (Experimental)
  Interventions: Biological: BMS-936558 (MDX-1106)

INTERVENTIONS:
Biological: BMS-936558 (MDX-1106) — Solution, Intravenous, 0.1 mg/kg - 10 mg/kg, Every 2 weeks, 3 years depending on response
  Other Names: BMS-936558
  Arms: Melanoma - BMS-936558 (MDX-1106)
Biological: BMS-936558 (MDX-1106) — Solution, Intravenous, 1 - 10 mg/kg, Every 2 weeks, 3 years depending on response
  Other Names: BMS-936558
  Arms: RCC - BMS-936558 (MDX-1106)
Biological: BMS-936558 (MDX-1106) — Solution, Intravenous, 10 mg/kg, Every 2 weeks, 3 years depending on response
  Other Names: BMS-936558
  Arms: mCRPC - BMS-936558 (MDX-1106)
Biological: BMS-936558 (MDX-1106) — Solution, Intravenous, 1 - 10 mg/kg, Every 2 weeks, 3 years depending on response
  Other Names: BMS-936558
  Arms: NSCLC - BMS-936558 (MDX-1106)
Biological: BMS-936558 (MDX-1106) — Solution, Intravenous, 10 mg/kg, Every 2 weeks, 3 years depending on response
  Other Names: BMS-936558
  Arms: CRC - BMS-936558 (MDX-1106)

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of MDX-1106 in patients with certain types of cancer. Another purpose is to determine how MDX-1106 is absorbed and distributed within the body, and how it's eventually eliminated.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Subjects must have mCRPC,RCC, MEL, Non-small-cell lung cancer (NSCLC), or Colorectal Cancer (CRC), that is advanced (non-resectable), or recurrent and for which no alternative, curative standard exists
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Must have at least 1 measurable lesion
* Subjects with mCRPC and with only non-measurable bone lesions must have either progression new lesions or have Prostate-specific antigen (PSA) progression within the 6-week period before study administration
* At least 1 and up to 5 prior systemic therapies for advanced/recurrent disease
* Prior treated brain or meningeal metastases must be without Magnetic resonance imaging (MRI) evidence of progression for at least 8 weeks and off immunosuppressive doses of systemic steroids for at least 2 weeks before study drug administration
* Prior systemic radiation therapy must have been completed at least 4 weeks before study drug administration. Prior focal radiotherapy completed at least 2 weeks prior to study drug administration
* Immunosuppressive doses of systemic medications, such as steroids or absorbed topical steroids must be discontinued at least 2 weeks before study drug administration
* Prior surgery that required general anesthesia must be completed at least 2 weeks before study drug administration. Surgery requiring local/epidural anesthesia must be completed at least 72 hours before study drug administration

Exclusion Criteria:

* History of severe hypersensitivity reactions to other Monoclonal antibody (mAb)s
* Subjects with any active autoimmune disease or a documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, except for subjects with vitiligo or resolved childhood asthma/atopy
* Prior therapy with an anti-Programmed death-1 (PD-1), anti-PD-L1, anti-PD-L2, or anti- Cytotoxic t-lymphocyte antigen-4 (CTLA-4) antibody (or any other antibody targeting T cell co-stimulation pathways)
* Known history of Human Immunodeficiency Virus
* Active infection requiring therapy, positive tests for Hepatitis B surface antigen or Hepatitis C ribonucleic acid (RNA)
* Underlying medical conditions that will make the administration of study drug hazardous
* Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids
* Use of other investigational drugs (drugs not marketed for any indication) within 28 days or at least 5 half-lives (whichever is longer) before study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2008-10-30 (Actual); Primary Completion 2013-02-04 (Actual); Study Completion 2020-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (13):
- United States (13):
  - Pinnacle Oncology Hematology, Scottsdale, Arizona
  - Yale University School Of Medicine, New Haven, Connecticut
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University Of Michigan Cancer Center, Ann Arbor, Michigan
  - Memorial Sloan Kettering Nassau, New York, New York
  - Carolina Biooncology Institute, Huntersville, North Carolina
  - Christ Hospital, Cincinnati, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Ctr, Nashville, Tennessee

REFERENCES:
- [Derived] Long GV, Larkin J, Schadendorf D, Grob JJ, Lao CD, Marquez-Rodas I, Wagstaff J, Lebbe C, Pigozzo J, Robert C, Ascierto PA, Atkinson V, Postow MA, Atkins MB, Sznol M, Callahan MK, Topalian SL, Sosman JA, Kotapati S, Thakkar PK, Ritchings C, Pe Benito M, Re S, Soleymani S, Hodi FS. Pooled Long-Term Outcomes With Nivolumab Plus Ipilimumab or Nivolumab Alone in Patients With Advanced Melanoma. J Clin Oncol. 2025 Mar 10;43(8):938-948. doi: 10.1200/JCO.24.00400. Epub 2024 Nov 6. PMID 39504507
- [Derived] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Drilon A, Wolchok JD, Carvajal RD, McHenry MB, Hosein F, Harbison CT, Grosso JF, Sznol M. Five-Year Survival and Correlates Among Patients With Advanced Melanoma, Renal Cell Carcinoma, or Non-Small Cell Lung Cancer Treated With Nivolumab. JAMA Oncol. 2019 Oct 1;5(10):1411-1420. doi: 10.1001/jamaoncol.2019.2187. PMID 31343665
- [Derived] Topalian SL, Sznol M, McDermott DF, Kluger HM, Carvajal RD, Sharfman WH, Brahmer JR, Lawrence DP, Atkins MB, Powderly JD, Leming PD, Lipson EJ, Puzanov I, Smith DC, Taube JM, Wigginton JM, Kollia GD, Gupta A, Pardoll DM, Sosman JA, Hodi FS. Survival, durable tumor remission, and long-term safety in patients with advanced melanoma receiving nivolumab. J Clin Oncol. 2014 Apr 1;32(10):1020-30. doi: 10.1200/JCO.2013.53.0105. Epub 2014 Mar 3. PMID 24590637
- [Derived] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 395 participants were enrolled and 306 were treated. 89 were not treated because they failed to meet study eligibility criteria or died prior to the initiation of treatment. All participants had received at least 1 prior cancer therapy. Study is on-going.
Groups:
- 0.1 mg/kg Nivolumab: 0.1 milligrams (mg) of nivolumab per kilogram (kg) of body weight (mg/kg)was administered intravenously (IV) every 2 weeks; Dosing on Days 1, 15, 29, and 43 (Cycle 1). Response was assessed between Days 52 and 56, before the first dose of the next cycle. Participants were treated until confirmed complete response (CR), worsening progressive disease (PD), or unacceptable toxicity, up to 12 cycles of treatment (96 weeks; 48 doses). Follow-up was up to 48 weeks. Re-initiation of study therapy was permitted for participants who entered the follow-up period with ongoing CR, partial response (PR), or stable disease (SD), who subsequently experienced confirmed PD.
- 0.3 mg/kg Nivolumab: 0.3 mg/kg nivolumab was administered by IV every 2 weeks; Dosing on Days 1, 15, 29, and 43 (Cycle 1). Response was assessed between Days 52 and 56, before the first dose of the next cycle. Participants were treated until confirmed CR, worsening PD, or unacceptable toxicity, up to 12 cycles of treatment (96 weeks; 48 doses). Follow-up was up to 48 weeks. Re-initiation of study therapy was permitted for participants who entered the follow-up period with ongoing CR, PR, or SD, who subsequently experienced confirmed PD.
- 1.0 mg/kg Nivolumab: 1.0 mg/kg nivolumab was administered by IV every 2 weeks; Dosing on Days 1, 15, 29, and 43 (Cycle 1). Response was assessed between Days 52 and 56, before the first dose of the next cycle. Participants were treated until confirmed CR, worsening PD, or unacceptable toxicity, up to 12 cycles of treatment (96 weeks; 48 doses). Follow-up was up to 48 weeks. Re-initiation of study therapy was permitted for participants who entered the follow-up period with ongoing CR, PR, or SD, who subsequently experienced confirmed PD.
- 3.0 mg/kg Nivolumab: 3.0 mg/kg nivolumab was administered by IV every 2 weeks; Dosing on Days 1, 15, 29, and 43 (Cycle 1). Response was assessed between Days 52 and 56, before the first dose of the next cycle. Participants were treated until confirmed CR, worsening PD, or unacceptable toxicity, up to 12 cycles of treatment (96 weeks; 48 doses). Follow-up was up to 48 weeks. Re-initiation of study therapy was permitted for participants who entered the follow-up period with ongoing CR, PR, or SD, who subsequently experienced confirmed PD.
- 10 mg/kg Nivolumab: 10 mg/kg nivolumab was administered by IV every 2 weeks; Dosing on Days 1, 15, 29, and 43 (Cycle 1). Response was assessed between Days 52 and 56, before the first dose of the next cycle. Participants were treated until confirmed CR, worsening PD, or unacceptable toxicity, up to 12 Cycles of treatment (96 weeks; 48 doses). Follow-up was up to 48 weeks. Re-initiation of study therapy was permitted for participants who entered the follow-up period with ongoing CR, PR, or SD, who subsequently experienced confirmed PD.
Period: Overall Study
Arm/Group | 0.1 mg/kg Nivolumab | 0.3 mg/kg Nivolumab | 1.0 mg/kg Nivolumab | 3.0 mg/kg Nivolumab | 10 mg/kg Nivolumab
Started | 17 | 18 | 86 | 54 | 131
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 17 | 18 | 86 | 54 | 131
Not completed — Adverse Event | 3 | 0 | 9 | 8 | 23
Not completed — Complete Response | 0 | 0 | 2 | 2 | 1
Not completed — Completed Maximum Cycles | 0 | 0 | 11 | 3 | 6
Not completed — Death | 0 | 0 | 0 | 0 | 2
Not completed — Disease Progression | 12 | 13 | 48 | 32 | 88
Not completed — non-specified | 0 | 0 | 4 | 2 | 3
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 6 | 3 | 4
Not completed — Treatment on-going | 2 | 5 | 5 | 4 | 4

BASELINE CHARACTERISTICS:
Population: All treated participants.
Groups:
- 0.1 mg/kg Nivolumab: Intravenous (IV) solution of 0.1 milligram nivolumab per kilogram of body weight (mg/kg) was administered every 2 weeks; Dosing on Days 1, 15, 29, and 43 of each treatment cycle.
- 0.3 mg/kg Nivolumab: 0.3 mg/kg nivolumab was administered every 2 weeks; Dosing on Days 1, 15, 29, and 43 of each treatment cycle.
- 1.0 mg/kg Nivolumab: 1.0 mg/kg nivolumab was administered every 2 weeks; Dosing on Days 1, 15, 29, and 43 of each treatment cycle.
- 3.0 mg/kg Nivolumab: 3.0 mg/kg nivolumab was administered every 2 weeks; Dosing on Days 1, 15, 29, and 43 of each treatment cycle.
- 10 mg/kg Nivolumab: 10 mg/kg nivolumab was administered every 2 weeks; Dosing on Days 1, 15, 29, and 43 of each treatment cycle.
- Total: Total of all reporting groups
Arm/Group | 0.1 mg/kg Nivolumab | 0.3 mg/kg Nivolumab | 1.0 mg/kg Nivolumab | 3.0 mg/kg Nivolumab | 10 mg/kg Nivolumab | Total
Number analyzed (Participants) | 17 | 18 | 86 | 54 | 131 | 306
Age, Continuous [Mean (Full Range); unit: years] | 57.5 [33 to 79] | 60.8 [29 to 85] | 61.8 [37 to 83] | 62.7 [32 to 81] | 63.1 [30 to 85] | 62.2 [29 to 85]
Age, Customized [Number; unit: participants]
  Less than (<) 65 years | 13 | 9 | 49 | 30 | 67 | 168
  Greater than or equal to (>)= 65 years | 4 | 9 | 37 | 24 | 64 | 138
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 26 | 21 | 43 | 103
  Male | 13 | 9 | 60 | 33 | 88 | 203
Tumor Type [Number; unit: participants]
  Squamous Non-Small Cell Lung Cancer (SQ NSCLC) | 0 | 0 | 15 | 18 | 21 | 54
  Non-Squamous NSCLC (NSQ NSCLC) | 0 | 0 | 18 | 19 | 37 | 74
  Melanoma | 17 | 18 | 35 | 17 | 20 | 107
  Renal Cell Carcinoma (RCC) | 0 | 0 | 18 | 0 | 16 | 34
  Castrate-Resistant Prostate Cancer (CRC) | 0 | 0 | 0 | 0 | 19 | 19
  MCRPC | 0 | 0 | 0 | 0 | 17 | 17
  NSCLC of Unspecified Histology | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Severe Adverse Events (AEs), Serious Adverse Events (SAEs), Treatment-Related AEs, Deaths, Discontinuation of Study Drug Due to AEs
Description: AE=any new unfavorable symptom, sign or disease or worsening of a preexisting condition that may not have a causal relationship with treatment.
  SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity or drug dependency/abuse; is life-threatening, an important medical event or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible or missing relationship to study drug. Death=during the study and up to 28 days past study discontinuation. The select AEs were determined using the Medical Dictionary for Regulatory Activities (MedDRA, v15.1) and graded using the Cancer Therapy Evaluation Program Common Terminology Criteria for Adverse Events (CTCAE), Version 3.0.
Time Frame: Day 1 to 70 days following last dose of study drug up to June 2013, approximately 4 years
Population: All participants who received at least 1 dose or any partial dose of nivolumab were analyzed.
Measure: Number; unit: participants
Arm/Group | 0.1 mg/kg Nivolumab | 0.3 mg/kg Nivolumab | 1.0 mg/kg Nivolumab | 3.0 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 17 | 18 | 86 | 54 | 131
participants
  SAE | 9 | 8 | 37 | 26 | 79
  Treatment-Related AE | 13 | 14 | 70 | 40 | 93
  All Deaths (within 100 days of last dose) | 4 | 4 | 18 | 9 | 40
  Treatment-Related Deaths | 0 | 0 | 1 | 0 | 1
  Discontinuation of Study Drug due to AEs | 3 | 0 | 12 | 12 | 30

2. Primary Outcome: Number of Participants With Abnormal Serum Chemistry Laboratory Values
Description: Alkaline phosphatase (ALP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Creatinine and Total Bilirubin. National Cancer Institute Common Terminology Criteria (CTC) version (v) 3.0 was used to determine Grade (Gr). Abnormal values for ALP, ALT and AST were based on grades; Gr 1: > 1.0 - 2.5 * upper limits of normal (ULN); Gr 2: > 2.5 - 5.0 * ULN; Gr 3: > 5.0 - 20.0 * ULN; Gr 4: > 20.0 * ULN. Abnormal values for Creatinine were based on Gr 1: > 1.0 - 1.5*ULN; Gr 2: > 1.5 - 3.0*ULN; Gr 3: > 3.0 - 6.0*ULN; Gr 4: > 6.0*ULN. Abnormal values for Total Bilirubin were based on Gr 1: > 1.0 - 1.5 * upper limits of normal (ULN); Gr 2: > 1.5 - 3.0 * ULN; Gr 3: > 3.0 - 10.0 * ULN; Gr 4: > 10.0 * ULN.
Time Frame: Day 1 up to June 2013, approximately 4 years
Population: All participants who received at least 1 dose or any partial dose of nivolumab who underwent the laboratory test.
Measure: Number; unit: participants
Arm/Group | 0.1 mg/kg Nivolumab | 0.3 mg/kg Nivolumab | 1.0 mg/kg Nivolumab | 3.0 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 17 | 18 | 86 | 54 | 131
participants
  ALP (Grades 1-2) | 8 | 7 | 21 | 11 | 38
  ALP (Grades 3-4) | 0 | 0 | 3 | 2 | 3
  ALT (Grades 1-2) | 6 | 3 | 25 | 13 | 18
  ALT (Grades 3-4) | 0 | 0 | 1 | 2 | 2
  AST (Grades 1-2) | 6 | 4 | 26 | 13 | 41
  AST (Grades 3-4) | 0 | 2 | 2 | 3 | 2
  Creatinine (Grades 1-2) | 5 | 9 | 21 | 9 | 34
  Creatinine (Grades 3-4) | 0 | 0 | 0 | 0 | 1
  Total Bilirubin (Grades 1-2) | 2 | 1 | 3 | 4 | 3
  Total Bilirubin (Grades 3-4) | 0 | 2 | 0 | 0 | 2

3. Secondary Outcome: Immunogenicity Assessment
Description: Classification of participants host immune response was based on the following definitions: Anti-Drug Antibody (ADA) Positive Subjects have with at least one ADA positive sample at any time after initiation of treatment. ADA positive subjects were further classified into categories with Persistent Positive defined as an ADA positive sample at 2 or more sequential timepoints at least 8 weeks apart.
Time Frame: Day 1 up to June 2013, approximately 4 years
Population: All participants who received at least 1 dose or any partial dose of nivolumab and were ADA-evaluable were analyzed.
Measure: Number; unit: participants
Arm/Group | 0.1 mg/kg Nivolumab | 0.3 mg/kg Nivolumab | 1.0 mg/kg Nivolumab | 3.0 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 14 | 14 | 66 | 46 | 103
participants
  ADA Positive | 6 | 2 | 7 | 2 | 4
  Persistant Positive | 1 | 0 | 1 | 0 | 0

4. Secondary Outcome: Objective Response Rate
Description: Tumor response was evaluated by the sponsor based on tumor assessments by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.0. Objective response rate (ORR) was defined as the proportion of participants who's confirmed best overall response (BOR) is either complete (CR) or partial (PR), where the denominator is the number of treated participants in the population of interest. Response was based on tumor measurements. Responders= complete response (CR) or partial response (PR). CR=disappearance of all target and non-target lesions; PR=at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the screening sum longest diameter. 95% Confidence intervals (CIs) were computed using the Clopper Pearson method.
Time Frame: Day 1 up to June 2013, approximately 4 years
Population: All participants who received at least 1 dose or any partial dose of nivolumab with an evaluable tumor response were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 0.1 mg/kg Nivolumab: Intravenous (IV) solution of 0.1 milligram nivolumab per kilogram of body weight (mg/kg) was administered every 2 weeks; Dosing on Days 1, 15, 29, and 43 (Cycle 1). Response was assessed between Days 52 and 56, before the first dose of the next cycle. Participants were treated until confirmed complete response (CR), worsening progressive disease (PD), or unacceptable toxicity, up to 12 Cycles of treatment (96 weeks; 48 doses). Follow-up was up to 48 weeks.
- 0.3 mg/kg Nivolumab: 0.3 mg/kg nivolumab was administered every 2 weeks; Dosing on Days 1, 15, 29, and 43 (Cycle 1). Response was assessed between Days 52 and 56, before the first dose of the next cycle. Participants were treated until confirmed CR, worsening PD, or unacceptable toxicity, up to 12 Cycles of treatment (96 weeks; 48 doses). Follow-up was up to 48 weeks.
- 1.0 mg/kg Nivolumab: 1.0 mg/kg nivolumab was administered every 2 weeks; Dosing on Days 1, 15, 29, and 43 (Cycle 1). Response was assessed between Days 52 and 56, before the first dose of the next cycle. Participants were treated until confirmed CR, worsening PD, or unacceptable toxicity, up to 12 Cycles of treatment (96 weeks; 48 doses). Follow-up was up to 48 weeks.
- 3.0 mg/kg Nivolumab: 3.0 mg/kg nivolumab was administered every 2 weeks; Dosing on Days 1, 15, 29, and 43 (Cycle 1). Response was assessed between Days 52 and 56, before the first dose of the next cycle. Participants were treated until confirmed CR, worsening PD, or unacceptable toxicity, up to 12 Cycles of treatment (96 weeks; 48 doses). Follow-up was up to 48 weeks.
- 10 mg/kg Nivolumab: 10 mg/kg nivolumab was administered every 2 weeks; Dosing on Days 1, 15, 29, and 43 (Cycle 1). Response was assessed between Days 52 and 56, before the first dose of the next cycle. Participants were treated until confirmed CR, worsening PD, or unacceptable toxicity, up to 12 Cycles of treatment (96 weeks; 48 doses). Follow-up was up to 48 weeks.
- All Dose Groups: All participants receiving Intravenous (IV) solution of 0.1-10 milligram nivolumab per kilogram of body weight (mg/kg) was administered every 2 weeks; Dosing on Days 1, 15, 29, and 43 (Cycle 1). Response was assessed between Days 52 and 56, before the first dose of the next cycle. Participants were treated until confirmed complete response (CR), worsening progressive disease (PD), or unacceptable toxicity, up to 12 Cycles of treatment (96 weeks; 48 doses). Follow-up was up to 48 weeks.
Arm/Group | 0.1 mg/kg Nivolumab | 0.3 mg/kg Nivolumab | 1.0 mg/kg Nivolumab | 3.0 mg/kg Nivolumab | 10 mg/kg Nivolumab | All Dose Groups
Number analyzed (Participants) | 17 | 18 | 35 | 37 | 59 | 129
percentage of participants
  SQ NSCLC (n=0,0,15,18,21,54) | 0 [NA to NA] — There are no participants so confidence interval was not calculated. | 0 [NA to NA] — There are no participants so confidence interval was not calculated. | 0 [NA to NA] — There are no participants so confidence interval was not calculated. | 22.2 [6.4 to 47.6] | 23.8 [8.2 to 47.2] | 16.7 [7.9 to 29.3]
  NSQ NSCLC (n=0,0,18,19,37,74) | 0 [NA to NA] — There are no participants so confidence interval was not calculated. | 0 [NA to NA] — There are no participants so confidence interval was not calculated. | 5.6 [0.1 to 27.3] | 26.3 [9.1 to 51.2] | 18.9 [8.0 to 35.2] | 17.6 [9.7 to 28.2]
  TOTAL NSCLC (n=0,0,33,37,59,129) | 0 [NA to NA] — There are no participants so confidence interval was not calculated. | 0 [NA to NA] — There are no participants so confidence interval was not calculated. | 3.0 [0.1 to 15.8] | 24.3 [11.8 to 41.2] | 20.3 [11.0 to 32.8] | 17.1 [11.0 to 24.7]
  Melanoma (n=17,18,35,17,20,107) | 35.3 [14.2 to 61.7] | 27.8 [9.7 to 53.5] | 31.4 [16.9 to 49.3] | 41.2 [18.4 to 67.1] | 20.0 [5.7 to 43.7] | 30.8 [22.3 to 40.5]
  Renal Cell Carcinoma (RCC) (n=0,0,18,0,16,34) | 0 [NA to NA] — There are no participants so confidence interval was not calculated. | 0 [NA to NA] — There are no participants so confidence interval was not calculated. | 27.8 [9.7 to 53.5] | 0 [NA to NA] — There are no participants so confidence interval was not calculated. | 31.3 [11.0 to 58.7] | 29.4 [15.1 to 47.5]

5. Secondary Outcome: Duration of Tumor Response
Description: Duration of tumor response (DOR) was calculated from the first date of response of complete response (CR) or partial response (PR) to the date of the first progressive disease (PD) or the date of death. Duration of response was censored at the last tumor assessment date if a responder did not have PD or death. Nonresponders were not included in the analysis. Median DOR was estimated by Kaplan-Meier analysis.
Time Frame: Day 1 up to June 2013, approximately 4 years
Population: All participants who received at least 1 dose or any partial dose of nivolumab with a measurable tumor response were analyzed.
Measure: Median (Full Range); unit: months
Arm/Group | 0.1 mg/kg Nivolumab | 0.3 mg/kg Nivolumab | 1.0 mg/kg Nivolumab | 3.0 mg/kg Nivolumab | 10 mg/kg Nivolumab | All Dose Groups
Number analyzed (Participants) | 17 | 18 | 35 | 37 | 59 | 129
months
  SQ NSCLC (n=0,0,15,18,21,54) | NA [NA to NA] — There are no participants in this group. | NA [NA to NA] — There are no participants in this group. | NA [NA to NA] — There are no participants with a response in this group. | NA [3.7 to 30.8] — Median duration of response has not been reached. | 19.1 [3.7 to 30.5] | NA [3.7 to 30.8] — Median duration of response has not been reached.
  NSQ NSCLC (n=0,0,18,19,37,74) | NA [NA to NA] — There are no participants in this group. | NA [NA to NA] — There are no participants in this group. | 14.7 [14.7 to 14.7] | 13.6 [5.6 to 17.0] | NA [1.4 to 22.7] — Median duration of response has not been reached. | 14.2 [1.4 to 22.7]
  All NSCLC (n=0,0,33,37,59,129) | NA [NA to NA] — There are no participants in this group. | NA [NA to NA] — There are no participants in this group. | 14.7 [14.7 to 14.7] | 17 [3.7 to 30.8] | 19.1 [1.4 to 30.5] | 17.0 [1.4 to 30.8]
  Mel (n=17,18,35,17,20,107) | NA [5.6 to 18.4] — Median duration of response has not been reached. | 20.7 [4.2 to 21.5] | 24.0 [3.9 to 24.9] | 17.5 [9.2 to 26.5] | 25.7 [17.0 to 26.9] | 22.9 [3.9 to 26.9]
  RCC (n=0,0,18,0,16,34) | NA [NA to NA] — There are no participants in this group. | NA [NA to NA] — There are no participants in this group. | 12.9 [9.2 to 17.5] | NA [NA to NA] — There are no participants in this group. | 12.9 [8.4 to 29.1] | 12.9 [8.4 to 29.1]

6. Secondary Outcome: Geometric Mean Maximum Serum Concentration (Cmax)
Description: Nivolumab in human serum was assayed by PPD® (Richmond, Virginia) using a cross-validated enzyme-linked immunosorbent assay (ELISA). Blood samples were assessed at all doses from a subset of participants. The pharmacokinetic (PK) parameter of Cmax was measured in micrograms per milliliter (µg/mL).
Time Frame: 1,4,8,24,48 and 96 hours post-dose timepoints on Day 1 of cycles 1 and 3
Population: All participants who received at least 1 dose or any partial dose of nivolumab and had adequate PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Groups:
- 0.1 mg/kg Nivolumab: Intravenous (IV) solution of 0.1 milligram nivolumab per kilogram of body weight (mg/kg) was administered every 2 weeks; Dosing on Days 1, 15, 29, and 43 of each cycle.
- 0.3 mg/kg Nivolumab: 0.3 mg/kg nivolumab was administered every 2 weeks; Dosing on Days 1, 15, 29, and 43 of each cycle.
- 1.0 mg/kg Nivolumab: 1.0 mg/kg nivolumab was administered every 2 weeks; Dosing on Days 1, 15, 29, and 43 of each cycle.
- 3.0 mg/kg Nivolumab: 3.0 mg/kg nivolumab was administered every 2 weeks; Dosing on Days 1, 15, 29, and 43 of each cycle.
- 10 mg/kg Nivolumab: 10 mg/kg nivolumab was administered every 2 weeks; Dosing on Days 1, 15, 29, and 43 of each cycle.
Arm/Group | 0.1 mg/kg Nivolumab | 0.3 mg/kg Nivolumab | 1.0 mg/kg Nivolumab | 3.0 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 15 | 17 | 17 | 13 | 14
micrograms per milliliter (µg/mL)
  Cycle 1/Day 1 (n=15,17,17,13,14) | 1.9 (23.6) | 7.0 (32.3) | 19.6 (29.5) | 61.3 (26.4) | 191.2 (40.0)
  Cycle 3/Day 1 (n=5,2,10,7,5) | 3.7 (42.2) | 17.8 (26.6) | 46.9 (26.1) | 132.0 (19.8) | 475.0 (24.6)

7. Primary Outcome: Number of Participants With Abnormal Hematology Laboratory Values
Description: Hemoglobin, Lymphocytes, Neutrophils, Platelets and Leukocytes. National Cancer Institute Common Terminology Criteria (CTC) version (v) 3.0 was used to determine Grade (Gr). Abnormal values for Hemoglobin were based on Gr 1: 10.0 - less than (<) lower limit of normal (LLN); Gr 2: 8.0 - < 10.0; Gr 3: 6.5 - < 8.0; Gr 4: < 6.5. Abnormal values for Lymphocytes were based on Gr 1: 0.8 - < 1.5; Gr 2: 0.5 - < 0.8; Gr 3): 0.2 - < 0.5; Gr 4: < 0.2. Abnormal values for Neutrophils were based on Gr 1: 1.5 - < 2.0; Gr 2: 1.0 - < 1.5; Gr 3: 0.5 - < 1.0; Gr 4: < 0.5. Abnormal values for Platelets were based on Gr 1: 75.0 - < lower limits of normal (LLN); Gr 2: 50.0 - < 75.0; Gr 3: 25.0 - < 50.0; Gr 4: < 25.0. Abnormal values for Leukocytes were based on Gr 1: 3.0 - < LLN; Gr 2: 2.0 - < 3.0; Gr 3: 1.0 - < 2.0; Gr4: < 1.0.
Time Frame: Day 1 up to June 2013, approximately 4 years
Population: All participants who received at least 1 dose or any partial dose of nivolumab who underwent the laboratory test.
Measure: Number; unit: participants
Arm/Group | 0.1 mg/kg Nivolumab | 0.3 mg/kg Nivolumab | 1.0 mg/kg Nivolumab | 3.0 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 17 | 18 | 86 | 54 | 131
participants
  Hemoglobin (Grades 1-2) | 12 | 12 | 58 | 46 | 101
  Hemoglobin (Grades 3-4) | 0 | 0 | 6 | 0 | 6
  Lymphocytes (Grades 1-2) | 9 | 15 | 64 | 43 | 101
  Lymphocytes (Grades 3-4) | 3 | 3 | 8 | 8 | 19
  Neutrophils (Grades 1-2) | 4 | 4 | 13 | 6 | 12
  Neutrophils (Grades 3-4) | 0 | 0 | 1 | 1 | 3
  Platelets (Grades 1-2) | 2 | 1 | 9 | 10 | 19
  Platelets (Grades 3-4) | 0 | 0 | 0 | 0 | 0
  Leukocytes (Grades 1-2) | 4 | 4 | 11 | 10 | 13
  Leukocytes (Grades 3-4) | 0 | 0 | 1 | 0 | 3

8. Secondary Outcome: Median Time of Maximum Serum Concentration (Tmax)
Description: Nivolumab in human serum was assayed by PPD® (Richmond, Virginia) using a cross-validated ELISA. Blood samples were assessed Blood samples were assessed at all doses from a subset of participants. The PK parameter of Tmax was measured in hours (h).
Time Frame: 1,4,8,24,48 and 96 hours post-dose timepoints on Day 1 of cycles 1 and 3
Population: All participants who received at least 1 dose or any partial dose of nivolumab and had adequate PK profiles.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | 0.1 mg/kg Nivolumab | 0.3 mg/kg Nivolumab | 1.0 mg/kg Nivolumab | 3.0 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 15 | 17 | 17 | 13 | 14
hours (h)
  Cycle 1/Day 1 (n=15,17,17,13,14) | 1.1 [0.3 to 51.0] | 1.2 [0.9 to 24.3] | 1.2 [0.9 to 48.0] | 2.1 [0.8 to 8.0] | 3.9 [1.0 to 48.2]
  Cycle 3/Day 1 (n=5,2,10,7,5) | 8.0 [0.6 to 24.0] | 24.7 [1.3 to 48.0] | 1.0 [0.9 to 24.1] | 4.0 [1.0 to 8.0] | 22.3 [1.0 to 24.5]

9. Secondary Outcome: Geometric Mean Area Under the Curve (AUC[TAU]) in One Dosing Interval Observed Post-Single Dose
Description: Nivolumab in human serum was assayed by PPD® (Richmond, Virginia) using a cross-validated ELISA. Blood samples were assessed at all doses from a subset of participants. The PK parameter of AUC was measured in micrograms*hours per milliliter (μg*h/mL).
Time Frame: 1,4,8,24,48 and 96 hours post-dose timepoints on Day 1 of cycles 1 and 3
Population: All participants who received at least 1 dose or any partial dose of nivolumab and had adequate PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hours per milliliter (μg*h/mL
Arm/Group | 0.1 mg/kg Nivolumab | 0.3 mg/kg Nivolumab | 1.0 mg/kg Nivolumab | 3.0 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 13 | 15 | 10 | 13 | 12
micrograms*hours per milliliter (μg*h/mL
  Cycle 1/Day 1 (n=13,15,10,13,12) | 279.4 (32.5) | 954.7 (26.9) | 3589.6 (23.8) | 8785.8 (22.7) | 31095.1 (25.4)
  Cycle 3/Day 1 (n=4,2,9,5,3) | 1101.4 (26.6) | 3406.1 (12.8) | 10190.4 (25.8) | 30640.3 (17.5) | 99621.7 (26.0)

10. Secondary Outcome: Geometric Mean Total Body Clearance of Drug From Serum (CLT)
Description: Nivolumab in human serum was assayed by PPD® (Richmond, Virginia) using a cross-validated ELISA. Blood samples Blood samples were assessed at all doses from a subset of participants. The PK parameter of CLT was measured in milliliters per hour (mL/h).
Time Frame: 1,4,8,24,48 and 96 hours post-dose timepoints on Day 1 of cycle 3
Population: All participants who received at least 1 dose or any partial dose of nivolumab and had adequate PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters per hour (mL/h)
Arm/Group | 0.1 mg/kg Nivolumab | 0.3 mg/kg Nivolumab | 1.0 mg/kg Nivolumab | 3.0 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 4 | 2 | 9 | 5 | 3
milliliters per hour (mL/h) | 8.3 (40.0) | 6.9 (17.8) | 8.0 (31.1) | 10.3 (18.1) | 8.5 (6.4)

11. Secondary Outcome: Mean Effective Half-life (T-HALFeff)
Description: Nivolumab in human serum was assayed by PPD® (Richmond, Virginia) using a cross-validated ELISA. Blood samples were assessed at all doses from a subset of participants. The PK parameter of T-HALFeff was measured in hours (h).
Time Frame: 1,4,8,24,48 and 96 hours post-dose timepoints on Day 1 of cycle 3
Population: All participants who received at least 1 dose or any partial dose of nivolumab and had adequate PK profiles.
Measure: Mean (Standard Deviation); unit: hours (h)
Arm/Group | 0.1 mg/kg Nivolumab | 0.3 mg/kg Nivolumab | 1.0 mg/kg Nivolumab | 3.0 mg/kg Nivolumab | 10 mg/kg Nivolumab
Number analyzed (Participants) | 4 | 2 | 9 | 5 | 3
hours (h) | 622 (235) | 555 (42) | 636 (267) | 661 (202) | 595 (80)

ADVERSE EVENTS:
Time Frame: Day 1 to 70 days following last dose of study drug up to February 2013
Description: Study initiated: October 2008; Primary endpoint: February 2013
Groups:
- 0.3 mg/kg Nivolumab: IV solution of 0.3 milligram nivolumab per kilogram of body weight (mg/kg) was administered every 2 weeks; Dosing on Days 1, 15, 29, and 43 of each treatment cycle.
- 1 mg/kg Nivolumab: IV solution of 1 milligram nivolumab per kilogram of body weight (mg/kg) was administered every 2 weeks; Dosing on Days 1, 15, 29, and 43 of each treatment cycle.
- 3 mg/kg Nivolumab: IV solution of 3 milligrams nivolumab per kilogram of body weight (mg/kg) was administered every 2 weeks; Dosing on Days 1, 15, 29, and 43 of each treatment cycle.
- 10 mg/kg Nivolumab: IV solution of 10 milligrams nivolumab per kilogram of body weight (mg/kg) was administered every 2 weeks; Dosing on Days 1, 15, 29, and 43 of each treatment cycle.
Arm/Group | 0.1 mg/kg Nivolumab | 0.3 mg/kg Nivolumab | 1 mg/kg Nivolumab | 3 mg/kg Nivolumab | 10 mg/kg Nivolumab
Serious Adverse Events (participants affected / at risk) | 9/17 | 8/18 | 37/86 | 26/54 | 79/131
Other Adverse Events (participants affected / at risk) | 17/17 | 17/18 | 83/86 | 51/54 | 130/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.1 mg/kg Nivolumab (N=17) | 0.3 mg/kg Nivolumab (N=18) | 1 mg/kg Nivolumab (N=86) | 3 mg/kg Nivolumab (N=54) | 10 mg/kg Nivolumab (N=131)
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Cranial nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 2 | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 2 | 1
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 1 | 0 | 3
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 3 | 1 | 4
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Urogenital haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Uveitis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 1 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 3 | 2 | 6
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1
Laryngeal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Metastases to penis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 2
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 6
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 2 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Lung infection pseudomonal (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Speech disorder (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 10
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 12 | 5 | 27
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 4
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Central nervous system haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 4
Intussusception (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Malignant soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 4 | 5
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 4 | 3 | 6
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Amylase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 2
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Gastrointestinal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 2
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 7
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Renal injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 5 | 2 | 19
Empyema (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 1
Hernia (General disorders) | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 2
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.1 mg/kg Nivolumab (N=17) | 0.3 mg/kg Nivolumab (N=18) | 1 mg/kg Nivolumab (N=86) | 3 mg/kg Nivolumab (N=54) | 10 mg/kg Nivolumab (N=131)
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 3 | 1 | 4
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 7 | 4 | 18
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 2 | 5
Candidiasis (Infections and infestations) | 1 | 1 | 0 | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 5 | 6
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 2 | 1 | 1
Depressed mood (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 13 | 5 | 12
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Eye pain (Eye disorders) | 1 | 0 | 0 | 2 | 0
Eyelid ptosis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 2 | 4 | 2 | 1
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 1 | 1
Hypertension (Vascular disorders) | 3 | 3 | 6 | 4 | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 5 | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 3 | 10 | 4 | 7
Hypothyroidism (Endocrine disorders) | 1 | 1 | 5 | 1 | 5
Insomnia (Psychiatric disorders) | 2 | 3 | 10 | 13 | 17
Leukopenia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 6 | 4 | 13
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 8 | 2 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 9 | 5 | 8
Neutrophil count increased (Investigations) | 2 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 1 | 4 | 3 | 8
Pain (General disorders) | 3 | 0 | 6 | 6 | 5
Proteinuria (Renal and urinary disorders) | 0 | 1 | 3 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 3 | 2 | 10
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0 | 0 | 1
Urogenital haemorrhage (Renal and urinary disorders) | 1 | 0 | 2 | 0 | 2
Vitiligo (Skin and subcutaneous tissue disorders) | 3 | 1 | 6 | 2 | 0
Weight increased (Investigations) | 0 | 1 | 5 | 5 | 5
Agitation (Psychiatric disorders) | 0 | 1 | 1 | 0 | 3
Ascites (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 2 | 1 | 2 | 3 | 4
Chills (General disorders) | 0 | 1 | 5 | 4 | 14
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 2 | 6 | 3 | 12
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 6 | 1 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 | 1 | 5
Flushing (Vascular disorders) | 1 | 1 | 3 | 4 | 4
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 4 | 5 | 13 | 12 | 24
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 2
Mental impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 3 | 2 | 6
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1 | 2 | 0 | 4
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 10
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 5 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 4 | 7
White blood cell count increased (Investigations) | 1 | 0 | 4 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 4 | 5 | 8
Anxiety (Psychiatric disorders) | 2 | 0 | 6 | 6 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 5 | 21 | 10 | 21
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatinine decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 4 | 2 | 6
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 2
Depression (Psychiatric disorders) | 1 | 1 | 6 | 5 | 9
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 37 | 23 | 36
Dry eye (Eye disorders) | 1 | 0 | 2 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 5 | 0 | 3
Fatigue (General disorders) | 10 | 8 | 42 | 31 | 75
Haematuria (Renal and urinary disorders) | 1 | 1 | 2 | 1 | 2
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0 | 2 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 1 | 18 | 4 | 10
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 1 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 7 | 1 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 4 | 3 | 6
Infusion site extravasation (General disorders) | 0 | 1 | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 5 | 3 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 1 | 1 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 2
Sensation of foreign body (General disorders) | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 5 | 0 | 8
Thyroxine free increased (Investigations) | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 1 | 2 | 4
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0
Visual impairment (Eye disorders) | 1 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 3 | 14 | 12 | 29
Weight decreased (Investigations) | 4 | 1 | 11 | 10 | 22
Xerosis (General disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 12 | 6 | 12
Axillary pain (General disorders) | 1 | 0 | 0 | 2 | 2
Blood glucose increased (Investigations) | 0 | 1 | 1 | 1 | 4
Brain oedema (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 3 | 0 | 9
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 7 | 6 | 31 | 17 | 46
Disease progression (General disorders) | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 1 | 4 | 5
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 1 | 6 | 7 | 16
Injection site discomfort (General disorders) | 1 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 7
Nodule (General disorders) | 2 | 0 | 1 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 10 | 7 | 15
Paraesthesia (Nervous system disorders) | 0 | 1 | 1 | 2 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 2 | 9
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 6 | 1 | 4
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 3
Viral infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 2 | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 2 | 4
Constipation (Gastrointestinal disorders) | 6 | 3 | 18 | 15 | 35
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 4 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 1 | 1
Dizziness (Nervous system disorders) | 3 | 4 | 15 | 9 | 25
Dry throat (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 5 | 9
Dysuria (Renal and urinary disorders) | 2 | 0 | 1 | 2 | 3
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Gait disturbance (General disorders) | 2 | 1 | 0 | 1 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 3
Granulocyte count decreased (Investigations) | 1 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 2 | 10
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 5 | 3 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 5 | 1
Melanosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 6 | 4 | 7
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 3 | 1 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 3 | 3 | 5
Prostatic specific antigen increased (Investigations) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 3 | 6 | 11 | 5 | 26
Rash (Skin and subcutaneous tissue disorders) | 3 | 5 | 27 | 13 | 25
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 3 | 7
Somnolence (Nervous system disorders) | 0 | 1 | 1 | 1 | 7
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 6 | 1 | 3
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 2 | 5 | 4 | 8
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 6 | 6 | 14
Asthenia (General disorders) | 0 | 0 | 6 | 2 | 10
Auriculotemporal syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 1 | 14 | 12 | 34
Blood testosterone decreased (Investigations) | 0 | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0 | 1
CD4 lymphocytes decreased (Investigations) | 1 | 0 | 0 | 1 | 3
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 6 | 4 | 12
Conjunctivitis (Eye disorders) | 0 | 1 | 1 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 0 | 7 | 1 | 17
Dysgeusia (Nervous system disorders) | 2 | 0 | 6 | 2 | 13
Facial wasting (Skin and subcutaneous tissue disorders) | 2 | 0 | 3 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2 | 8 | 2 | 4
Lacrimation increased (Eye disorders) | 0 | 1 | 3 | 2 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 11 | 6 | 23
Nausea (Gastrointestinal disorders) | 2 | 4 | 22 | 17 | 39
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 1 | 0 | 2
Oedema peripheral (General disorders) | 4 | 2 | 18 | 9 | 24
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | 5 | 12
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 4 | 0
Sunburn (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 3 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 0 | 6
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 2 | 3 | 5
Alanine aminotransferase increased (Investigations) | 0 | 1 | 11 | 2 | 6
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 3 | 2 | 6
Blood uric acid increased (Investigations) | 0 | 0 | 3 | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 21 | 17 | 42
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 22 | 17 | 25
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 2
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Genital erythema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 0 | 3
Haemoglobin decreased (Investigations) | 2 | 3 | 12 | 7 | 18
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 4 | 5 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 4 | 3 | 3
Influenza like illness (General disorders) | 2 | 1 | 6 | 3 | 2
Macular degeneration (Eye disorders) | 1 | 0 | 0 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Mucous stools (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 3 | 14
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 1 | 2 | 2 | 4
Oral herpes (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 4 | 21 | 8 | 20
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 5 | 6 | 3 | 13
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 9 | 2 | 3
Blood phosphorus decreased (Investigations) | 0 | 0 | 1 | 0 | 7
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 1 | 5 | 10
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 4 | 4 | 15
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3 | 8
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2
Haemorrhage (Vascular disorders) | 0 | 1 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 5 | 0 | 4
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 1
Lentigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 2 | 3 | 4 | 5 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 3 | 7
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2 | 2 | 7
Otitis media (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 6 | 7
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 1 | 5
Rhinitis (Infections and infestations) | 1 | 1 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 1 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1 | 2
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Thyroxine free decreased (Investigations) | 1 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 2 | 2 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 2 | 0 | 4 | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trials primary publication.